CLINICAL TRIAL: NCT06972368
Title: Efficacy Study of Enhanced Home-Based Transcranial Direct Current Stimulation (tDCS) on Depressive Symptoms in Borderline Personality Disorder (BPD): A Pilot Randomized Controlled Trial
Brief Title: Home-Based tDCS for Depression in BPD
Acronym: TENTADIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-4050
Record Dates: First submitted 2025-04-22; First posted 2025-05-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder (MDD); Borderline Personality Disorders
Keywords: Neuromodulation; personality; tDCS; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Borderline Personality Disorder; Depression | interventions — Transcranial Direct Current Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tDCS (Experimental): 14 sessions of active tDCS, twice daily, each lasting 30 minutes and separated by an interval of minimum at 2 hours. Ideally, sessions will be scheduled at the same time each day.
  Interventions: Device: tDCS; Procedure: Treatment as Usual (TAU); Procedure: Psychoeducation
- Sham tDCS (Placebo Comparator): 14 sessions of sham tDCS, twice daily, each lasting 30 minutes and separated by an interval of minimum at 2 hours. Ideally, sessions will be scheduled at the same time each day.
  Interventions: Procedure: Treatment as Usual (TAU); Procedure: Psychoeducation; Device: Sham-tDCS

INTERVENTIONS:
Device: tDCS — Description:
  Participants randomized to this arm will receive 14 sessions of home-based transcranial Direct Current Stimulation (tDCS), administered twice daily for 30 minutes over 7 consecutive days. Each session will use a 2mA current with a SNAPstrap™ montage targeting the left dorsolateral prefrontal cortex (F3) with the anode and the right DLPFC (F4) with the cathode. Sessions include a 30-second ramp-up and ramp-down. The total delivered charge will be 48 coulombs.
  Enhancement component:
  Each session will be paired with cognitive and emotional enhancement strategies:
  Emotion regulation script (DBT-inspired, personalized and pre-written based on a moderately dysregulated situation).
  Cognitive training via Lumosity, targeting executive functions and memory.
  Arms: tDCS
Procedure: Treatment as Usual (TAU) — Description:
  Throughout the study, participants are required to maintain stable pharmacological and psychotherapeutic regimens, defined as:
  No changes in medications or therapy for at least 6 weeks after tDCS initiation.
  TAU is provided by participants' regular treating physician or mental health professional, independent of the study team.
  TAU includes psychotropic medication, psychotherapy, and case management, as clinically indicated.
Procedure: Psychoeducation — All participants receive access to a structured online psychoeducation program before randomization.
  This includes:
  * Short videos (8-14 minutes each) covering BPD, depression, neuromodulation, therapeutic success factors, and tDCS.
  * Multiple-choice quizzes (MCQs) to ensure comprehension.
  * Delivered in French with English subtitles. Designed to improve understanding of BPD and associated treatments, including the rationale for tDCS.
Device: Sham-tDCS — Description:
  Participants randomized to this arm will receive 14 sessions of sham tDCS, with identical scheduling and device setup as the active condition. The session mimics real tDCS (same SNAPstrap montage, ramp-up and ramp-down of 30 seconds), but no current is delivered after the initial 30 seconds.
  Enhancement component:
  Participants follow the same emotional regulation script and Lumosity cognitive training during
  Arms: Sham tDCS

SUMMARY:
The present study aims to assess the feasibility of home-based tDCS in remote and urban areas (primary objective).

The secondary aim is to obtain a preliminary assessment of the efficacy of 14 home-based tDCS sessions in reducing depressive symptoms in BPD patients with moderate to severe depressive episodes and BPD symptoms.

Exploratory objectives include assessing the impact on neuropsychological and psychosocial functioning, anxiety, physical activity, sleep disorders, and addiction.

Additionally, we aim to investigate the sociodemographic and clinical factors that are linked to the most favorable response to tDCS in addressing both depressive and BPD symptoms.

We also aim to assess the feasibility of using a smartwatch as an outcome measure in this population.

Finally, we intend to gather preliminary data on the effectiveness of an online psychoeducational program specifically designed for patients with BPD.

Researchers will compare active tDCS to sham tDCS to see if active treatment is more effective in treating depression in this population.

Participants will:

* Receive 14 sessions of either active or sham tDCS over one week, delivered at home
* Complete psychological and neurocognitive assessments at baseline, post-treatment, and at 6 weeks
* Wear actigraphy monitors and complete questionnaires to assess sleep, physical activity, and other mental health outcomes

This trial will also explore the feasibility of delivering tDCS in both urban and rural settings.

DETAILED DESCRIPTION:
Abstract Background Depressive disorders are the most common comorbidity among individuals with Borderline Personality Disorder (BPD), affecting over 85% of patients and leading to high recurrence rates and resistance to treatment. Traditional pharmacological and psychotherapeutic interventions often show limited efficacy in this population, highlighting the need for innovative treatment strategies. Emerging evidence suggests that the dorsolateral prefrontal cortex (DLPFC) plays a crucial role in the pathophysiology of both Major Depressive Disorder (MDD) and BPD. In addition, non-invasive brain stimulation, particularly transcranial Direct Current Stimulation (tDCS), has shown promising results in alleviating depression and improving BPD symptoms when targeting the DLPFC. The development of home-based tDCS presents new opportunities for accessible and cost-effective interventions. However, no study has specifically investigated its effects on MDD in the context of BPD.

Methods This double-blind randomized controlled trial (RCT) will assess the efficacy of home-based tDCS in reducing depressive symptoms in BPD patients who are experiencing moderate to severe depressive episodes. A total of 60 participants will be randomly assigned to either active or sham tDCS for 14 sessions over two weeks. The primary outcome is the remission rate according to the Montgomery-Åsberg Depression Rating Scale (MADRS) scores six weeks after treatment initiation. Secondary outcomes include changes in BPD symptom severity, anxiety, sleep quality, and functional impairment. Exploratory analyses will evaluate the impact of tDCS on neuropsychological functioning, physical activity, and addiction. Sociodemographic variables will be considered in predicting treatment response. Feasibility and acceptability outcomes will also be assessed, including patient adherence and satisfaction (visual analog score). All assessments will be conducted at baseline, post-treatment, and during follow-ups up to three months after treatment ends.

Discussion The findings will address both the clinical efficacy and feasibility of tDCS in real-world settings, contributing to the development of scalable neuromodulation strategies for individuals with BPD and comorbid depression.

ELIGIBILITY:
Inclusion Criteria:

1. To be aged between 18 and 65.
2. To meet the DSM-IV criteria for BPD.
3. To present a moderate depressive episode, defined as a MADRS score ≥ 20 (V1 and V3).
4. To be capable to consent to participate in the study.
5. To speak either French or English.
6. Participants must have a prescribing doctor or mental health professional responsible
7. To maintain a stable psychopharmacological and psychotherapeutic intervention.
8. To have access to internet an a smartphone.
9. To demonstrate proficiency in independently using a tDCS device.
10. To be able to pick up and return the remote tDCS device.

Exclusion Criteria:

- 1. To have a history of Epilepsy. 2. To have a contraindication for tDCS Medical Devices. 3. To have a history of Cerebrovascular Surgery. 4. To present scalp Conditions Affecting tDCS Electrode Placement. 5. To have a history of bipolar disorder. 6. To present social or medical conditions limiting the autonomous use of remote tDCS.

7. To be pregnant. 8. To be currently undergoing neuromodulation treatment. 9. To be currently using benzodiazepines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline (Day 0), Week 1 (Day 7), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Month 3; primary endpoint at Week 6 after initial stimulation.
  The MADRS is a clinician-administered scale with ten items designed to assess the severity of depressive symptoms. Each item is scored from 0 to 6, yielding a total score ranging from 0 to 60 (higher is more severe). The assessment requires approximately 15 to 20 minutes to complete. It possesses high internal consistency, evidenced by a Cronbach's alpha of 0.85-0.89, and demonstrates sensitivity to change, making it suitable for evaluating treatment efficacy. The scale has been validated in French and can be administered over the phone.

SECONDARY OUTCOMES:
Borderline Symptom List (BSL-23) | Baseline (Day 0), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  The BSL-23 is a 23-item self-report questionnaire designed to assess the severity of BPD symptoms over the past week (higher scores indicate more severe symptoms). This shortened version of the BSL-95 is widely used for routine monitoring of BPD. The assessment takes approximately 10 minutes to complete. The BSL-23 demonstrates excellent internal consistency, with a Cronbach's alpha of roughly .94 for the French version.
Quick Inventory of Depressive Symptomatology (QIDS) | Baseline (Day 0), Week 1 (Day 7), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  Quick Inventory of Depressive Symptomatology (QIDS): The QIDS is a 16-item self-report questionnaire based on DSM-IV criteria for major depression. It assesses symptom severity over the past 7 days (higher is more severe) and takes approximately 5 to 10 minutes to complete. The assessment has good internal consistency, with a Cronbach's alpha of 0.69 to 0.89 (75). It has been translated into French.
Borderline Personality Disorder Severity Index (BPDSI) | Pre-intervention (immediately prior to tDCS/sham) and Month 3.
  The BPDSI is a 70-item semi-structured interview designed to assess the frequency and severity of BPD symptoms over the past three months. It captures critical symptoms and behaviours associated with BPD, such as self-harm, emotional dysregulation, and interpersonal conflicts. The interview takes approximately 45 to 60 minutes to complete. The BPDSI yields highly reliable (ICC = .93) and internally consistent (Cronbach's α = .85) scores. The BPDSI has been translated into French and used in clinical research, although its psychometric properties have not yet been validated for the French version.
Personality Disorder Severity Scale (PDS-ICD-11) | Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham).
  The PDS-ICD-11 is a clinician-rated instrument designed to assess the severity of personality disorder features by the International Classification of Diseases, 11th Revision (ICD-11). This scale evaluates impairments in self-functioning (identity and self-direction) and interpersonal functioning (empathy and intimacy), the core components of personality pathology defined by the ICD-11 framework. The PDS-ICD-11 provides a dimensional assessment, categorizing severity into five levels: no personality dysfunction, personality difficulty, mild personality disorder, moderate personality disorder, and severe personality disorder. This nuanced approach allows for a standardized and comprehensive evaluation of personality dysfunction, facilitating both diagnosis and the monitoring of treatment outcomes. A version has been translated into French.
Barratt Impulsiveness Scale (BIS-11) | Baseline (Day 0), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  The BIS is a 30-item self-report questionnaire that evaluates various dimensions of impulsivity, including attentional, motor, and non-planning impulsivity. It takes approximately 10 minutes to complete. The BIS has good internal consistency, with a Cronbach's alpha ranging from 0.69 to 0.83, indicating satisfactory scale homogeneity. A French version is available.
World Health Organization Disability Assessment Schedule (WHODAS 2.0, 12-item version) | Baseline (Day 0), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  The WHODAS 2.0 (12-item) is a brief self-report questionnaire designed to assess disability and functioning across six domains: cognition, mobility, self-care, getting along with others, life activities, and participation in society. Higher scores indicate greater functional impairment. Developed by the World Health Organization, it has good internal consistency, with a Cronbach's alpha ranging from 0.87 to 0.94, indicating excellent scale homogeneity. The scale is available in French (85)and English and takes approximately 5-10 minutes to complete.
Beck Anxiety Inventory (BAI) | Baseline (Day 0), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  The BAI is a 21-item self-report questionnaire designed to assess the severity of anxiety symptoms experienced over the past week. The items focus on physical symptoms of anxiety, such as nervousness and heart palpitations. The BAI takes approximately 10 minutes to complete. It has excellent internal consistency, with a Cronbach's alpha of 0.91.
Antidepressant Treatment History Form - Short Form (ATHF-SF) | Baseline.
  The ATHF-SF is a clinician-administered tool designed to assess a patient's history of antidepressant treatments systematically. It provides a concise and structured way to document the type, dosage, duration, and adequacy of antidepressant trials and the patient's response to these treatments. The ATHF-SF helps determine the extent of previous antidepressant exposure and can identify potential treatment-resistant depression. It will enable us to classify patients into five stages, from no treatment to ECT.
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Baseline (Day 0), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  ASSIST is a widely used tool developed by the World Health Organization (WHO) for the screening and measurement of addiction across various substances, including alcohol, tobacco, cannabis, and opioids. ASSIST is designed for use in clinical and research settings to assess both current and lifetime use, and associated risks of substance use disorders. The tool consists of eight questions that measure the frequency of use, cravings, and negative impacts of substances on physical, mental, social, and legal aspects of the individual's life, allowing for a quick and comprehensive screening. Psychometric evaluations of ASSIST demonstrate high reliability and validity across various settings and populations. Studies report good internal consistency, with Cronbach's alpha values ranging from 0.80 to 0.88 and high test-retest reliability (ICC = 0.90), indicating consistent results over time.
Pittsburg Sleep Questionnaire Inventory (PSQI) | This assessment will be administered at multiple time points: inclusion, pre-randomization, immediately after tDCS or sham stimulation, six weeks post-stimulation, and three months post-stimulation.
  The PSQI is a 19-item self-report questionnaire designed to assess subjective sleep quality across seven components, including sleep latency, duration, sleep disturbances, and daytime dysfunction. Higher scores indicate poorer sleep quality. The PSQI takes approximately 10 minutes to complete. It has good internal consistency, with a fair or reasonable Cronbach's alpha coefficient (ranging from 0.64 to 0.83. The instrument has been validated in French.
Psychophysiological parameters | The wristwatch will be worn starting from the second visit-one week after inclusion-until just after the tDCS or sham-tDCS session, two weeks later.
  In this study, participants will wear FitBit watches to objectively measure several key outcomes related to sleep, physical activity, and physiological metrics. Sleep data will include the total sleep duration and the time spent in each stage (light, deep, and REM sleep). Physical activity will be assessed by tracking the number of steps taken per day and the number of active minutes. Additionally, the investigators will monitor physiological activity, focusing on heart rate variability (HRV) and heart rate (HR) frequency, providing insights into participants' cardiovascular and autonomic functioning.
The Personality Inventory for DSM-5 (PID-5) | Baseline (Day 0), Pre-intervention (immediately prior to first tDCS/sham), Post-intervention (within 1 day after of tDCS/sham), Week 6 and Month 3.
  The PID-5 is a validated psychometric tool designed to assess maladaptive personality traits described in the DSM-5 Alternative Model for Personality Disorders. In clinical research, the PID-5 is an outcome measure by capturing dimensional traits across five broad domains: Negative Affectivity, Detachment, Antagonism, Disinhibition, and Psychoticism. Each domain consists of more specific facets that provide a detailed profile of personality pathology. Using the PID-5, researchers can quantify changes in these traits over time, making it a valuable tool for evaluating the effectiveness of therapeutic interventions. Additionally, its use in cross-sectional and longitudinal studies allows for assessing personality trait stability or improvement following treatment.
N-back task | This assessment will be administered at two time points: one week after inclusion and immediately after the tDCS or sham stimulation.
  The N-back task is designed to evaluate working memory and will be administered online. Participants will view a sequence of stimuli and indicate when the current stimulus matches one presented "n" steps earlier. The task duration is typically 15-20 minutes, depending on the difficulty level (e.g., 2-back or 3-back).
Go/No-Go | This assessment will be administered at two time points: one week after inclusion and immediately after the tDCS or sham stimulation.
  The Go/No-Go task measures impulsivity and inhibitory control. Participants respond to "go" stimuli while inhibiting responses to "no-go" stimuli. This task generally takes around 10 minutes to complete. These assessments are integrated into the protocol to evaluate key cognitive domains (planning, working memory, and inhibitory control). They will be conducted remotely, ensuring accessibility and participant convenience while collecting valid and reliable data.

CONTACTS AND LOCATIONS:
Locations (1):
- IUSMM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Description:
  De-identified individual participant data (IPD) underlying published results will be made available to qualified researchers upon reasonable request. Data will include clinical assessments, questionnaire scores, and tDCS usage logs. No personal identifiers will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available 12 months after publication of the main results and for a period of 5 years.
Access Criteria: Researchers must submit a methodologically sound proposal describing the purpose of the data use. Requests will be reviewed by the study's principal investigator and data access committee. A data-sharing agreement will be required.